CLINICAL TRIAL: NCT01154491
Title: Multicenter Double-bind Randomized Trial of Ferric Carboxymaltose With or Without Erythropoietin for the Prevention of Red-cell Transfusion in Hip Fracture Perioperative Period.
Brief Title: Efficacy of Ferric Carboxymaltose With or Without EPO Reducing Red-cell Transfusion Packs in Hip Fracture Perioperative Period
Acronym: PAHFRAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Maximo Bernabeu Wittel, Maximo Bernabeu Wittel, Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAHFRAC-01; 2009-015865-30 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-07-01 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Hip Fractures
Keywords: hip fractures; blood substitutes; blood transfusion; intravenous infusion; erythropoietin, recombinant; frail elderly
MeSH Terms: conditions — Hip Fractures | interventions — ferric carboxymaltose; Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Two placebos: placebo for ferric carboxymaltose and placebo for erythropoietin
  Interventions: Drug: Placebo
- FE (Experimental): Ferric carboxymaltose and placebo for erythropoietin
  Interventions: Drug: Ferric carboxymaltose
- EPOFE (Experimental): Ferric carboxymaltose and erythropoietin
  Interventions: Drug: Ferric carboxymaltose; Drug: Erythropoietin

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferinject®: Ferric carboxymaltose: 2 vials of 10 mL containing each 500 mg iron, diluted in 250 mL normal saline for injection. Study drug to be administered by infusion immediately after preparation.
  Placebo for erythropoietin: 1 mL normal saline for subcutaneous injection.
  Other Names: Intravenous iron
  Arms: EPOFE; FE
Drug: Erythropoietin — Erythropoetin: 40,000 units subcutaneous (unique dose).
  Other Names: EPO
  Arms: EPOFE
Drug: Placebo — Placebo for ferric carboxymaltose: 250 mL normal saline for intravenous administration.
  Placebo for erythropoietin: 1 mL normal saline for subcutaneous injection.
  Arms: Placebo

SUMMARY:
In order to evaluate the efficacy of ferric carboxymaltose + erythropoietin versus ferric carboxymaltose versus placebo in reducing the percentage of patients who receive red-cell transfusion in the perioperative period of hip fracture, a multicenter, randomized, parallel groups, double-blind clinical trial in adult patients admitted for osteoporotic hip fracture is designed. Required sample size is of 87 patients per arm (87x3 = 261). Primary efficacy variable is the percentage of patients who receive red-cell transfusion during hospitalization; secondary end-points: average red-cell packs per patient,haemoglobin at 24 h and 72h after the intervention, at the time of hospital discharge and 60 days after hospital discharge, hospital stay and mortality during hospital-stay and 60 days afterwards. Adverse clinical events and side effects are assessed as safety variables. In addition health related quality of life will be measured at inclusion and after 60 days. A cost-efficacy analysis (by means of incremental cost-efficacy method using as a primary endpoint each patient not requiring transfusion, and as secondary end-point every patient who survived the index admission is performed). The investigators would like to demonstrate a double benefits: optimizing precious resource such as blood products and reducing complications arising from their use.

DETAILED DESCRIPTION:
Three arms of treatments: A: ferric carboxymaltose and erythropoietin, B: ferric carboxymaltose and placebo, arm C: two placebos. Primary objective:reduction of red-cell packs needed for elderly patients with osteoporotic hip fracture which requires surgical intervention in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years and older.
* Osteoporotic hip fracture which require surgical intervention
* Haemoglobin levels between 90-120 g/L
* Signed informed consent form

Exclusion Criteria:

* Bone marrow diseases which could interfere in the erythropoietic process (acute or chronic myelodysplastic syndromes or myeloproliferative diseases, and/or infiltration of the bone marrow due to solid or lymphatic neoplasms)
* Blood coagulation diseases or currently treated with oral anticoagulants and/or heparin at therapeutic doses.
* Documented allergy and/or previous intolerance and/or contraindication of erythropoietin use and/or intravenous iron.
* Patients with rheumatoid arthritis and/or another demonstrated origin of inflammatory anemia and/or not controlled arterial hypertension.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 303 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Reduce red-cell transfusion packs | 60 days after hospital discharge
  percentage of patients who receive red-cell transfusion during hospitalization

SECONDARY OUTCOMES:
Average red-cell packs per patient | end of study
Haemoglobin level | 24 h and 72h after the intervention, at the time of hospital discharge and 60 days after hospital discharge
Number of hospitalization days | end of study
  number of days inhospital
Death rate with all causes mortality | end of study
Adverse Events | end of study
  adverse clinical events, side effects, Serious Adverse Events (SAE) and Suspected Unexpected Serious Adverse Reaction(SUSAR)
Quality of life | end of study
  health related quality of life
cost-efficacy analysis | end of study
  means of incremental cost-efficacy method (using as a primary endpoint each patient not requiring transfusion, and as secondary end-point every patient who survived the index admission)

CONTACTS AND LOCATIONS:
Overall Officials: Máximo Bernabeu-Wittel, MD, Principal Investigator — Hospital Universitario Virgen del Rocio. Sevilla
Locations (14):
- Spain (14):
  - Hospital Universitario de Albacete, Albacete, Albacete
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de la Vega Baja, Orihuela, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville, España
  - Hospital Donostia, San Sebastián, Guipúzcoa
  - Hospital Infanta Elena, Huelva, Huelva
  - Hospital Lucus Augusti, Lugo, Lugo
  - Hospital de la Serranía de Ronda, Ronda, Malaga
  - Hospital Comarcal de la Axarquía, Vélez-Málaga, Málaga
  - Hospital San Juan de Dios del Aljarafe, Bormujos, Sevilla
  - Hospital Universitario Virgen Macarena, Seville, Seville
  - Hospital Universitario Río Hortega, Valladolid

REFERENCES:
- [Derived] Bernabeu-Wittel M, Romero M, Ollero-Baturone M, Aparicio R, Murcia-Zaragoza J, Rincon-Gomez M, Monte-Secades R, Melero-Bascones M, Rosso CM, Ruiz-Cantero A; PAHFRAC-01 Investigators. Ferric carboxymaltose with or without erythropoietin in anemic patients with hip fracture: a randomized clinical trial. Transfusion. 2016 Sep;56(9):2199-211. doi: 10.1111/trf.13624. Epub 2016 May 14. PMID 27195774
- [Derived] Bernabeu-Wittel M, Aparicio R, Romero M, Murcia-Zaragoza J, Monte-Secades R, Rosso C, Montero A, Ruiz-Cantero A, Melero-Bascones M; PAHFRAC-01 investigators. Ferric carboxymaltose with or without erythropoietin for the prevention of red-cell transfusions in the perioperative period of osteoporotic hip fractures: a randomized contolled trial. The PAHFRAC-01 project. BMC Musculoskelet Disord. 2012 Feb 21;13:27. doi: 10.1186/1471-2474-13-27. PMID 22353604